CLINICAL TRIAL: NCT03561584
Title: A Randomized, Placebo-controlled Pilot Study of Sulfasalazine for the Treatment of Primary Sclerosing Cholangitis (PSC)
Brief Title: Sulfasalazine for the Treatment of Primary Sclerosing Cholangitis
Acronym: SHIP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua Korzenik, Director, Crohn's and Colitis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P000019
Record Dates: First submitted 2018-05-14; First posted 2018-06-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-12

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Sclerosing; Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangitis | interventions — Sulfasalazine

STUDY DESIGN:
Intervention Model Description: There are two arms in this trial: active drug and placebo. We are recruiting remotely throughout the United States so an individual anywhere in the US with PSC and IBD can be enrolled.
Who Masked: Participant, Care Provider
Masking Description: Participants and Providers will be masked until Week 14. If a subject continues past week 14, the study becomes Open-Label and participants are given the option to continue on the active drug for an additional 8 weeks. We are recruiting remotely throughout the United States so an individual anywhere in the US with PSC and IBD can be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Drug (Sulfasalazine) (Active Comparator)
  Interventions: Drug: Sulfasalazine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulfasalazine — Patients will be initiated on a low dose of sulfasalazine (500 mg) twice daily (bid). Dosage will be increased throughout the study.
  Other Names: Azulfidine
  Arms: Active Drug (Sulfasalazine)
Drug: Placebo — Patients will be initiated on 1 placebo tablet twice daily (bid). Dosage will be increased throughout the study.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blinded placebo controlled trial to assess the benefit of sulfasalazine in the treatment of PSC. The specific objectives of this study are to determine if sulfasalazine treatment 1) results in reduced serum ALP and other biomarkers of liver injury in PSC; 2) improves PSC patient symptoms; and 3) is safe in patients with PSC.

We are recruiting remotely throughout the United States so an individual anywhere in the US with PSC and IBD can be enrolled.

DETAILED DESCRIPTION:
As there is a strong association between PSC and IBD, it is reasonable to hypothesize that a therapy of proven benefit for UC may prove to also be effective for PSC. Unfortunately, several therapies which are indicated for the treatment of UC have not been effective in PSC including anti-TNF therapies and other anti-inflammatory medications. Sulfasalazine and mesalamine, medications commonly used for the treatment of UC, may be exceptions to this trend. While this therapy has never been formally tested in PSC, some retrospective reports suggest a possible benefit. Our current understanding of the mechanism of action of these medications suggests there is reasonable to believe they may also be effective in PSC.

We are recruiting remotely throughout the United States so an individual anywhere in the US with PSC and IBD can be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-80
2. A diagnosis of PSC for at least 6 months based upon cholangiography (ERCP or MRCP) demonstrating intrahepatic and/or extrahepatic biliary strictures, beading or irregularity consistent with PSC.
3. ALP > 1.67 times the upper limit of normal (ULN) at screening
4. Inflammatory bowel disease
5. Subject must either be on a stable dose of ursodeoxycholic acid for > 6 months prior to screening or have been discontinued > 4 weeks prior to screening (enrollment of patients who are on UDCA will be limited to 50% of all enrolled patients).

We are recruiting remotely throughout the United States so an individual anywhere in the US with PSC and IBD can be enrolled.

Exclusion Criteria:

1. Anticipated need for liver transplant within one year as determined by Mayo PSC risk score treatment
2. Evidence of decompensated liver disease such as variceal bleeding, ascites, or hepatic encephalopathy.
3. Evidence of advanced liver disease including MELD score > 10, bilirubin > 3.0, platelet count < 100,000; or INR > 1.4
4. Concomitant chronic liver disease including alcohol related liver disease, chronic hepatitis B or C infection, haemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency, non-alcoholic steatohepatitis, autoimmune hepatitis, or primary biliary cholangitis
5. Secondary causes of sclerosing cholangitis
6. Known intolerance to sulfasalazine (including but not limited to allergy to sulfa or mesalamine) or folic acid
7. History of cholangiocarcinoma or colon cancer within 5 years
8. History of colectomy with > 1/3 bowel resected
9. Treatment with any investigational agents, within two months or 5 half-lives of the investigational product, whichever is longer.
10. Active illicit drug or alcohol abuse
11. Current or past use of sulfasalazine within 6 months of enrollment.
12. Need for chronic use of antibiotics
13. Evidence of bacterial cholangitis within 6 months of enrollment
14. In patients with Ulcerative Colitis, simple clinical colitis activity index of > 4 or, if Crohn's disease, a Harvey-Bradshaw index of > 5
15. Chronic kidney injury (eGFR < 59)
16. Pregnancy or lactation

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Mean Alkaline Phosphatase (ALP) | Baseline through the end of the Study at Week 22
  Proportion of patients with reduction of mean ALP < 1.5 x ULN at end of treatment
Normalization of ALP below the upper limit of normal | Baseline through the end of the Study at Week 22
  Assessment in number of patients whose ALP normalizes

SECONDARY OUTCOMES:
Overall changes in ALP levels | Baseline through the end of the Study at Week 22
  Proportion of patients with ALP > or < 1.5 x ULN at end of treatment
Changes in blood tests | Baseline through the end of the Study at Week 22
  Change in mean Liver Function Tests (e.g. Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), total bilirubin) and C-reactive Protein
Adverse Events | Baseline through the end of the Study at Week 22
  Unexpected and Serious Adverse Events will be examined
Changes in Mayo PSC risk score | Baseline through the end of the Study at Week 22
  Number of patients with changes in Mayo PSC risk score
Changes in Modified Fatigue Scale (MFS) | Baseline through the end of the Study at Week 22
  Number of patients with changes in MFS score
Changes in pruritus visual analog scale (VAS) | Baseline through the end of the Study at Week 22
  Number of patients with changes in VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Korzenik, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No